CLINICAL TRIAL: NCT07156929
Title: Kinetics and Metabolism of Nicotinamide Provided as a Dietary Supplementation: CICR-NAM as Food for Special Medicinal Purposes (FSMP)
Brief Title: Kinetics and Metabolism of Nicotinamide Provided as a Dietary Supplementation
Acronym: CICR-NAM_PK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D 417/24
Record Dates: First submitted 2025-07-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Infection (for Example, Pneumonia, Bronchitis); Respiratory Infection Virus; Community Acquired Pneumonia (CAP); COPD Acute Exacerbation; Inflammatory Bowel Disease (IBD)
Keywords: Nicotinamide; Controlled-Ileocolonic-Release Nicotinamide; CICR-NAM; Community Acquired Pneumonia; COPD; Inflammatory Bowel Disease; Crohn; Colitis
MeSH Terms: conditions — Respiratory Tract Infections; Pneumonia; Bronchitis; Community-Acquired Pneumonia; Inflammatory Bowel Diseases; Pulmonary Disease, Chronic Obstructive; Colitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 500 mg/d CICR-NAM (Active Comparator): 500 mg/d controlled-ileocolonic-release nicotinamide for 28 d
  Interventions: Dietary Supplement: Controlled-ileocolonic-release nicotinamide (CICR-NAM): 500 mg/d
- 1000 mg/d CICR-NAM (Active Comparator): 500 mg/d controlled-ileocolonic-release nicotinamide for 28 d
  Interventions: Dietary Supplement: Controlled-ileocolonic-release nicotinamide (CICR-NAM): 1000 mg/d

INTERVENTIONS:
Dietary Supplement: Controlled-ileocolonic-release nicotinamide (CICR-NAM): 500 mg/d — Controlled-ileocolonic-release nicotinamide (CICR-NAM) film-coated tablets release 500 mg nicotinamide per tablet at a pH of 7, leading to a delayed and prolonged systemic exposure to nicotinamide and to exposure of the ileum and colon including the gut microbiome.
  Arms: 500 mg/d CICR-NAM
Dietary Supplement: Controlled-ileocolonic-release nicotinamide (CICR-NAM): 1000 mg/d — Controlled-ileocolonic-release nicotinamide (CICR-NAM) film-coated tablets release 500 mg nicotinamide per tablet at a pH of 7, leading to a delayed and prolonged systemic exposure to nicotinamide and to exposure of the ileum and colon including the gut microbiome.
  Arms: 1000 mg/d CICR-NAM

SUMMARY:
The diet of patients with reduced tryptophan serum levels that are either hospitalized for acute respiratory infection or treated for chronic inflammatory diseases such as inflammatory bowel diseases (in- or outpatients) is supplemented with controlled-ileocolonic-release nicotinamide (CICR-NAM) at doses of 500 mg or 1000 mg per day for four weeks. In the COVit-2 trial (NCT04751604), nicotinamide supplementation including CICR-NAM has been shown to accelerate physical recovery from mild-to-moderate COVID-19 (for publication, see References). The main objective of this open-label case series is to investigate the pharmacokinetics and metabolism of nicotinamide in patients with more severe respiratory infections or chronic inflammatory conditions. In addition, patients can optionally provide information on their quality of life and fatigue status.

ELIGIBILITY:
Inclusion Criteria:

* Serum tryptophan levels below normal range.
* Acute, infectious respiratory disease requiring treatment (e.g. proven acute SARS-CoV-2 or influenza virus infection with inpatient treatment) or chronic inflammatory disease (e.g. chronic inflammatory bowel disease) in remission or in acute relapse (outpatient or inpatient treatment).

Exclusion Criteria:

* Inability to give informed consent.
* Pregnancy or breastfeeding.
* Serious other illness, e.g. cancer.
* Anemia: Hb <10 mg/dL.
* Intake of medication to raise the pH value in the stomach (e.g. proton pump inhibitors, H2 receptor antagonists or antacids) in higher doses over a longer period of time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-04-20 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in plasma concentrations of nicotinamide (NAM) and its main metabolites N-methylnicotinamide (NMN) and N-methyl-2-pyridone-5-carboxamide (2-Py) as well as nicotinic acid (NA) and nicotinuric acid (NUA) | From baseline (day 1) until day 2 (minimum), day 3 or day 8
  Simultaneous measurement by liquid chromatography with tandem mass spectrometry.

SECONDARY OUTCOMES:
Changes in serum concentrations of tryptophan and its metabolites | From baseline (day 1) until day 2 (minimum), day 3 or day 8
  Simultaneous measurement by liquid chromatography with tandem mass spectrometry.
Changes in quality of life (EuroQoL 5 Dimensions 5 Levels [EQ-5D-5L] questionnaire; optional) | Weekly from baseline until week 4
  The EQ-5D-5L health states can be summarised using a 5-digit code representing the 5 dimensions 'mobility', 'self-care', 'activity', 'pain' and 'anxiety' with 5 levels each from 1 = no problem to 5 = maximum problem. In addition, the subjects report their overall self-perceived health-related quality of life using the Visual Analogue Scale (VAS) from 0 = worst health one can imagine to 100 = best health one can imagine.
Changes in fatigue (Functional Assessment of Chronic Illness Therapy - Fatigue [FACIT-F] questionnaire; optional) | Weekly from baseline until week 4
  The FACIT-F questionnaire is a 40-item measure that assesses self-reported fatigue and its impact upon daily activities and function. The higher the subscores and total score, the better the self-perceived quality of life (for the total score, the range is from 0 to 160).

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Schreiber, Prof. Dr. Dr. h.c., Principal Investigator — University Hospital Schleswig-Holstein; Jan Heyckendorf, Prof. Dr., Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- University Hospital Schleswig-Holstein, Campus Kiel, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: Yes
Specific requests by academic researchers can be addressed to the principal investigators. On the basis of such a request including a detailed analysis plan, access might be provided, subject to a decision of the Ethics Committee of the Medical Faculty of Kiel University to ensure compliance with privacy laws, data protection and requirements for consent and anonymization.

REFERENCES:
- [Background] Schreiber S, Waetzig GH, Lopez-Agudelo VA, Geisler C, Schlicht K, Franzenburg S, di Giuseppe R, Pape D, Bahmer T, Krawczak M, Kokott E, Penninger JM, Harzer O, Kramer J, von Schrenck T, Sommer F, Zacharias HU; COVit-2 Study Group; Millet Pascual-Leone B, Forslund SK, Heyckendorf J, Aden K, Hollweck R, Laudes M, Rosenstiel P. Nicotinamide modulates gut microbial metabolic potential and accelerates recovery in mild-to-moderate COVID-19. Nat Metab. 2025 Jun;7(6):1136-1149. doi: 10.1038/s42255-025-01290-1. Epub 2025 May 12. PMID 40355744